CLINICAL TRIAL: NCT03999112
Title: A Case Series Examination of Metacognitive Reflection and Insight Therapy (MERIT) on Individual Negative Symptoms of Schizophrenia
Brief Title: Effect of Metacognitive Therapy on Negative Symptoms: a Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GN19MH107
Record Dates: First submitted 2019-05-20; First posted 2019-06-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Schizophrenia
Keywords: psychological therapy; metacognitive reflection
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Single case experimental design (SCED). Participants will be randomised to a baseline period, and after either 4, 6 or 8 weeks they will then be allocated to the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metacognitive Reflection and Insight Therapy (MERIT) 4 week (Experimental): Standard MERIT + 4 week baseline period
  Interventions: Other: Metacognitive Reflection and Insight Therapy (MERIT)
- Metacognitive Reflection and Insight Therapy (MERIT) 6 week (Experimental): Standard MERIT + 6 week baseline period
  Interventions: Other: Metacognitive Reflection and Insight Therapy (MERIT)
- Metacognitive Reflection and Insight Therapy (MERIT) 8 week (Experimental): Standard MERIT + 8 week baseline period
  Interventions: Other: Metacognitive Reflection and Insight Therapy (MERIT)

INTERVENTIONS:
Other: Metacognitive Reflection and Insight Therapy (MERIT) — A psychological therapy aiming to increase the ability of individuals to synthesise perceptions about themselves and others; to then form complex narratives which recognise the occurrence of these within particular social contexts; and to use these to form responses to psychological problems.

SUMMARY:
Negative symptoms (e.g. diminished pleasure and motivation) are common in people with a diagnosis of schizophrenia. Little is known about the psychological mechanisms involved in negative symptom development and maintenance and there is limited evidence for current treatment options. Some research suggests that difficulties with metacognition; the capacity to develop and use complex ideas about oneself and others, may predict experiences of negative symptoms. This study will investigate whether Metacognitive Reflection and Insight Therapy (MERIT) improves metacognition in people experiencing negative symptoms, and if metacognitive changes lead to observable differences in behavioural manifestations of negative symptoms (e.g. low activity levels).

Data will be collected via standardised assessments of metacognition and negative symptoms. Activity levels will be measured with actigraphy, which has been shown to capture differential activity patterns for individuals who experience negative symptoms compared to control groups. An assessment will also be made of whether improvements in specific aspects of metacognition (e.g. self-reflectivity) relate to changes in individual negative symptoms, such as motivation levels, and other markers of personal change, including personal and social performance, insight, and beliefs about recovery.

Additionally, factors that may have impacted on the study results, such as therapist adherence to the treatment, will be reported. Eligible patients with capacity to consent will be recruited from the inpatient rehabilitation psychology services in National Health Service (NHS) Greater Glasgow and Clyde. They will be aged 18 or over, have a schizophrenia spectrum disorder diagnosis, and experience current negative symptoms. The target sample size is up to 8 patients. Participants will be measured at baseline and will receive up to 26 sessions of the MERIT treatment approach. Any therapeutic change will be observed via changes from assessments at baseline to the assessments in the initial, middle and last therapy sessions, and also metacognitive assessments at two other randomly selected time-points during therapy.

DETAILED DESCRIPTION:
Hypotheses around metacognitive changes:

It is hypothesised that metacognition scores on the Metacognition Assessment Scale - Abbreviated (MAS-A) will increase with the implementation of Metacognitive Reflection and Insight Therapy (MERIT) over the course of treatment. It is also estimated that this will be related to changes in therapist-rated metacognition, and measures of participant insight (using the Beck Cognitive Insight Scale; BCIS). It is also anticipated that changes in participants' metacognition will also be related to whether therapist metacognition appears to match the level of participant metacognition demonstrated within session.

Hypotheses around impact on negative symptoms and secondary outcomes:

It is estimated that fewer manifestations of negative symptoms (e.g. low-activity levels) will be observed over the course of therapy compared to the baseline period, and that this will also be related to changes in the Clinical Assessment Interview of Negative Symptoms (CAINS), the Self-experience of Negative Symptoms scale (SNS), the Personal and Social Performance Scale (PSP), the Personal Questionnaire: Rapid Scaling Technique (PQRST) and the Questionnaire about the Process of Recovery (QPR).

Design rationale:

The SCED methodology and the use of measures of metacognition and negative symptoms over time was chosen because this allows examination of they key study hypotheses without the need for a standard control group design. This, coupled with the use of standardised measures, ensures that researchers can be confident that any therapeutic changes demonstrated in the study are more likely to be attributed to MERIT than by chance. This also serves as a cost-effective option for investigating the relationship between metacognition and negative symptoms and will identify ways MERIT can be tailored to these specific symptoms, giving an evidence base to build upon and understand how these factors, and particularly their subdomains, are related.

Timeline:

Training of therapists in MERIT has taken place. Recruitment will begin once ethical approval is in place. Participants will be randomly allocated to a baseline period of 4, 6, or 8 weeks during which they will complete a baseline assessment and receive instruction on how to use the actigraph device, and data on all measures other than the MAS-A and the PQRST (which are in-session data), will be recorded during the baseline period. The intervention will last up to 26 sessions, with interpretation, analyses and write up of the research completed thereafter. To avoid the introduction of bias to subsequent assessments or the intervention itself, there will be no interim analyses of the results, however researchers and therapists will remain vigilant to any detrimental affects to participants and any desire participants may have to stop participating in the research.

Additionally, the researcher will have no discussions with the therapists about how therapy is progressing for any participants, unless there is significant risk to the participant or others. Both MERIT sessions and the assessments by the researcher will take place in rehab wards in NHS Greater Glasgow and Clyde (GG&C).

Procedure:

Participants will be subject to researcher assessment (in scoring of the the CAINS and the MAS-A) and also therapist rated metacognition, and the PSP which is based on key worker observations. Participants medical access will also be accessed proportionately to gain demographic information and information about diagnosis. Participants will be made aware of this at the point of providing informed consent, and any perceived risk to the participant or others that is identified during these observations will be discussed with the participant where appropriate. Additionally, participants will provide self-report information via their report of time use and answers on the BCIS, SNS, the PQRST, and the QPR and to demographic questions. Also participants will be asked to wear actigraph devices which will allow participants' activity levels to be tracked. Participants will again be informed of the purposes of collecting these data and any concerns participants have will be discussed throughout the study as required. Whether participants continue to provide consent will also be checked throughout the study and participants will be able to stop providing data on a particular measure alone, or discontinue the study entirely, if they no longer consent to this.

The target sample size will be up to 8 participants, this has previously been identified as sufficient for SCED methodology, and given that participants will be identified through rehab wards in NHS GG&C, it is anticipated that this target sample size can be met.

Feasibility:

It is anticipated that inclusion criteria for this research will ensure individuals eligible will be those who experience persistent negative symptoms and who are already be expected to receive some form of psychological therapy as part of their NHS care and treatment. Therefore, the testing of MERIT, which is aimed at the treatment of negative symptoms, while novel, should not incur any additional cost or NHS resources.

ELIGIBILITY:
Inclusion Criteria:

* Receiving inpatient rehabilitation services in NHS GG&C
* Schizophrenia spectrum diagnosis, defined by diagnostic codes F20-29 from the International Classification of Diseases - 10th Edition (ICD-10; World Health Organization, 1992)
* Sufficient capacity to provide informed consent, as determined by treating clinician
* Score 4 or above from a possible total score of 8 in any subdomain of negative symptoms (alogia, avolition,anhedonia, social withdrawal or diminished emotional range) on the Self-evaluation of Negative Symptoms measure (SNS)
* Moderate to severe scores on either the motivation and pleasure scale or the expression scale of the Clinical Assessment Interview for Negative Symptoms (CAINS; resulting in a required score of 18 or above for items 1-9 and a score of 8 or above for items 10-13)

Exclusion Criteria:

* None, assuming all Inclusion Criteria are met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in Negative symptoms | Between baseline and week 1/week 13/week 26 of intervention
  Activity levels as measured by actigraphy device

SECONDARY OUTCOMES:
Clinical Assessment Interview for Negative Symptoms | baseline and week 1, week 13 and week 26 of intervention
  Clinical interview measuring 13 items on a scale of 0 - 4 where 0 indicates no impairment, 1 indicates mild deficit, 2 indicates moderate deficit, 3 indicates moderately severe deficit, and 4 indicates severe deficits. Items are summed and form a total score and 2 subscale scores on the motivation and pleasure and also the expression subscale. A greater score indicates greater negative symptom impairments.
Self-Evaluation of Negative Symptoms | baseline and week 1, week 13 and week 26 of intervention
  20 items measuring negative symptoms rated by participant on a likert scale where 0 represents strongly disagree, 1 represents somewhat agree, and 2 represents strongly agree. Total score is the sum of all items and a greater score indicates greater levels of negative symptoms.
Metacognition Assessment Scale - Adapted | baseline and week 1, week 13 and week 26 of intervention, plus two randomly selected timepoints between weeks 1-13 of intervention and weeks 14-26 of intervention.
  4 components of metacognition rated from rater assessment of participant interviews - self-reflectivity, understanding the mind of the other, decentration, mastery. Ratings on a scale of 0-1 for each level of metacognition demonstrated in each subscale with half a point awarded when partially demonstrated. Ranges for subscales are: self-reflectivity, 0-9; understanding the mind of the other, 0-7; decentration, 0-3; and mastery, 0-9. Total score is the sum of all subscales and ranges from 0-28. For all scores a lower score indicates lower levels of metacognition.
Metacognition Assessment Scale - Adapted, therapist rated | measured on a weekly basis during intervention period (up to 26 weeks)
  4 components of metacognition rated by therapist based on therapy session - self-reflectivity, understanding the mind of the other, decentration, mastery. Ratings on a scale of 0-1 for each level of metacognition demonstrated in each subscale with half a point awarded when partially demonstrated. Ranges for subscales are: self-reflectivity, 0-9; understanding the mind of the other, 0-7; decentration, 0-3; and mastery, 0-9. Total score is the sum of all subscales and ranges from 0-28. For all scores a lower score indicates lower levels of metacognition.
Beck Cognitive Insight Scale | baseline and week 1, week 13 and week 26 of intervention
  15 items measuring cognitive insight separated into two subscales: self-reflectiveness and self-certainty. Participants will rate items between 0-3, resulting in a total score of between 0 and 27 for the self-reflectiveness subscale and 0 - 18 for the self-certainty subscale. For both subscales, higher scores are reflective of higher self-reflectiveness and higher self-certainty. The two scales are compared by calculating a composite index, which is the sum of self-reflectivity minus the sum of self-certainty subscales.
Personal and Social Performance scale | baseline and week 1, week 13 and week 26 of intervention
  Measure giving an impression of social interactions, personal care, and aggression or disturbing behaviours exhibited. 4 domains of functioning (socially useful activities, including work or academic study; personal and social relationships; self-care; and disturbing and aggressive behaviours) are rated by a key worker from the following ordinal options: absent, mild, manifest, marked, severe and very severe. The number of difficulties across four areas and their severity are used to select a score between 1-100 at a 10 point interval and clinical judgement is used to adjust the score within the 10 point interval by accounting for other areas of social functioning. Participants thus receive a score between 1 and 100.
Personal Questionnaire Rapid Scaling Technique | measured on a weekly basis during intervention period (up to 26 weeks)
  1-5 meaningful personal statements agreed between participant and therapist; presented and asked if intensity greater or less than previous discussion. All items scored between 1-5 as a likert scale for the following 5 ordinal options: not at all (1), occasionally (2), sometimes (3), often (4), most of the time (5). A greater score indicates an item is a greater problem for participant than a lower score. Items are not aggregated.
Time Use Survey | baseline and week 1, week 13 and week 26 of intervention
  A measure of time use based on participant report of activities across a given week. Descriptive characteristics of activities are recorded including whether this was with other individuals, whether the activity was someone else's idea, whether these activities were started recently or the participant intends to take up new activities, and how satisfied the participant is with their overall levels of activity on a likert scale from 1-5 where 1 indicates very satisfied, 2 somewhat satisfied, 3 neither satisfied or dissatisfied, 4 somewhat dissatisfied, and 5 very dissatisfied. Activities are scored against criteria ranging from 0-4 where a lower score indicates a lower activity level and level of independence. Sum scores are reported for number of activities, activity level according to criteria, number of activities with others, new activities and satisfaction with activities.
Questionnaire about the Process of Recovery | baseline and week 1, week 13 and week 26 of intervention
  15 items about the process of recovery rated by participants where items are selected from the following ordinal responses: disagree strongly, disagree, neither agree nor disagree, agree and agree strongly. Each of these responses represent a score of 0-4 respectively, and the total score is a summation of scores for all items. A higher score represents more experiences of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Hamish McLeod, PhD CPsychol, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No